CLINICAL TRIAL: NCT02245997
Title: Local Control With Reduced-dose Radiotherapy for High-Risk Neuroblastoma
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-186
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Last update posted 2025-09-29 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma
Keywords: Reduced-dose Radiotherapy; 14-186
MeSH Terms: conditions — Neuroblastoma

ARMS (1):
- patients with high-risk neuroblastoma (Experimental): Patients undergo external beam radiation therapy using IMRT or proton beam RT twice daily for 5-6 weekdays (10-12 treatments). Patients will be evaluated by physical exams, CT scan or MRI of the primary site, and MIBG at, 6, 12, 18 and 24 months (+/- 6 weeks).
  Interventions: Radiation: External beam radiotherapy; Radiation: proton beam RT

INTERVENTIONS:
Radiation: External beam radiotherapy
  Other Names: IMRT
Radiation: proton beam RT

SUMMARY:
The purpose of this study is to give 12T a smaller dose of radiation in order to decrease these late side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of neuroblastoma (International Classification of Disease for Oncology [ICD-O] morphology 9500/3) confirmed by MSKCC pathologic review
* Patients must have high-risk neuroblastoma as defined by the COG Risk Stratification Schema

  o Patients with International agreement on staging (INSS) stage 4 are eligible with the following:
* MYCN amplification, regardless of age or additional biologic features
* Age >18 months, regardless of biologic features OR
* Age 1-18 months, with any of the 3 following unfavorable biologic OR features: MYCN amplification, unfavorable pathology, and/or DNA index = 1

  o Patients with INSS stage 3 are eligible with the following:
* MYCN amplification, regardless of age or additional biologic features OR
* Age > 18 months with unfavorable pathology, regardless of MYCN status

  o Patients with INSS stage 2a or 2b are eligible with the following:
* MYCN amplification, regardless of age or additional biologic features

  o Patients with INSS stage 4s are eligible with the following:
* MYCN amplification, regardless of additional biologic features Patients must have undergone chemotherapy and surgery for high-risk neuroblastoma prior to enrollment on trial.
* Age at time of enrollment of ≥1 month and ≤18 years
* Female patients of childbearing potential must have a negative pregnancy test within 14 days of radiation start.
* Female patients who are lactating must agree to stop breast-feeding.
* Sexually active patients of childbearing potential must agree to use effective contraception.

Exclusion Criteria:

* Patients with gross residual tumor after surgical resection
* Patients who have received prior radiotherapy at or adjacent to the primary tumor bed
* Patients with any concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make them inappropriate candidates for entry into this study.

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2014-09; Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
assess local control rates treatment response | 3 yeas
  will be assessed via imaging (CT+/- MRI and MIBG) and clinical evidence at the primary site post completion of treatment. The baseline scan will be the pre-irradiation CT scan. Local failure is defined as a relapse in the primary tumor bed or adjacent lymph nodes.

SECONDARY OUTCOMES:
event-free survival | 3 years
  will be performed for each patient using clinical data and imaging. Events are defined as failure (loco-regional and/or distant), treatment-related malignancy, or death.
Assessment of toxicity | 3 years
  will occur at the pre-specified follow-up time-points using the CTCAE version 4.0 grading system.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Wolden, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/